CLINICAL TRIAL: NCT07306715
Title: Comparison of Pectopexy Operations With and Without Mesh Use After Laparoscopic Hysterectomy for Pelvic Organ Prolapse.
Brief Title: Laparoscopic Pectopexy With and Without Mesh Use for Pelvic Organ Prolapse.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Şener Gezer, Şener Gezer, MD, Associate Prof., Principal Investigator, Kocaeli University, School of Medicine, Department of Obstetrics and Gynecology, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAEK/18.bI.02
Record Dates: First submitted 2025-12-14; First posted 2025-12-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Genital Prolapse
Keywords: pectopexy; mesh
MeSH Terms: interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Pectopexy without mesh (Experimental): In this group of patients, the Laparoscopic Pectopexy operation will be performed without the use of mesh material after hysterectomy. Not using mesh will be protective against possible erosion reactions that may develop in the postoperative period. Laparoscopic hysterectomy is performed using the standard procedure with a uterine manipulator; after sealing the uterine arteries, the vagina is cut at the level of the uterine manipulator cuff and sutured. The vaginal cuff will be fixed to the pectineal ligament with No. 1, non-absorbable Prolene suture.
  Interventions: Procedure: Meshless Laparoscopic Pectopexy
- Laparoscopic Pectopexy with mesh (Active Comparator): In this group of patients, the Laparoscopic Pectopexy operation will be performed using mesh material after hysterectomy. Laparoscopic hysterectomy is performed using the standard procedure with a uterine manipulator; after sealing the uterine arteries, the vagina is cut at the level of the uterine manipulator cuff and sutured. The vaginal cuff will be fixed to the pectineal ligament with polypropylene mesh.
  Interventions: Procedure: Laparoscopic Pectopexy with mesh

INTERVENTIONS:
Procedure: Meshless Laparoscopic Pectopexy — The vaginal cuff will be fixed to the pectineal ligament with No. 1, non-absorbable Prolene suture.
  Arms: Laparoscopic Pectopexy without mesh
Procedure: Laparoscopic Pectopexy with mesh — The vaginal cuff will be fixed to the pectineal ligament with polypropylene mesh.
  Arms: Laparoscopic Pectopexy with mesh

SUMMARY:
Genital apical prolapse refers to the descent of the vaginal apex, uterus, or cervix, and surgical treatment is required for adequate apical support. Laparoscopic pectopexy is a surgical method developed as an alternative to the gold standard, sacrocolpopexy, in the treatment of genital organ prolapse, especially for obese patients for whom dissection is difficult. The vaginal cuff is attached to the pectineal ligament with polypropylene mesh in the standard technique. The use of mesh is subject to serious restrictions due to complications such as mesh erosion. Surgical methods without using a mesh may be safer treatment options for patients with genital prolapse. This study aimed to compare the results of Laparoscopic Pectopexy surgery with and without the use of mesh material after hysterectomy.

DETAILED DESCRIPTION:
After ethics committee approval, patients with stage 2 and above pelvic organ prolapse according to the POP-Q staging system, who have completed their fertile period and do not want uterus preservation, will be included in the study. The stage of prolapse according to POP-Q and other gynecological examination findings will be recorded at the initial examination. Prolapse and its impact on the quality of life will be recorded preoperatively and 12 months postoperatively with the Prolapse Quality of Life Questionnaire (P-QOL). Patients will be called for examination 12 months after the operation. The ratio of women with stage 2 or greater vaginal cuff prolapse according to the Pelvic Organ Prolapse Quantification (POP-Q) system is the main outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients older than 40 years and younger than 80 years old with symptomatic uterine prolapse
* Patients who provided written consent for the surgical procedure
* Patients who do not wish to preserve their uterus

Exclusion Criteria:

* Patients who cannot obtain anesthesia approval for laparoscopic surgery
* Patients who have a confirmed or suspected pregnancy
* Patients who have abnormal uterine/cervical/vaginal bleeding
* Patients with biopsy-confirmed endometrial hyperplasia or cervical dysplasia
* Patients with pathology-confirmed genital cancer
* Patients undergone chemotherapy or radiotherapy for any type of cancer

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with symptomatic uterine prolapse
Enrollment: 60 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Apical descensus relapse rate | 12 months after surgery
  The ratio of women with stage 2 or greater vaginal cuff prolapse according to the Pelvic Organ Prolapse Quantification (POP-Q) system.

SECONDARY OUTCOMES:
Prolapse Quality of Life (P-QOL) | Preoperative day and 12 months after surgery
  The questionnaire has nine items, each of which has a 4-point scoring system and a total score of 0-100. A high total score indicates worsening of the quality of life of women with pelvic organ prolapse.

OTHER OUTCOMES:
De novo central or lateral defect cystocele rate | 12 months after surgery
  The ratio of women with stage 2 or greater central or lateral defect cystocele according to the Pelvic Organ Prolapse Quantification (POP-Q) system
De novo rectocele rate | 12 months after surgery
  The ratio of women with stage 2 or greater rectocele according to the Pelvic Organ Prolapse Quantification (POP-Q) system

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Bıyık, M.D., Study Chair — Kütahya Sağlık Bilimleri University
Locations (1):
- Kocaeli University, School of Medicine, Köseköy, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erdem B, Salman S, Usta ZK, Bacak HB, Ozkan MD, Ceken AT, Isik EY, Kumbasar S, Gencer FK, Baghaki HS, Kacar T, Aslan GN, Bulut B. A Novel Approach for Apical Prolapse Surgery: Meshless Pectopexy (Salman's Modification). Int Urogynecol J. 2025 Aug;36(8):1701-1705. doi: 10.1007/s00192-025-06107-z. Epub 2025 Apr 1. PMID 40167602
- [Background] Aleksandrov A, Smith AV, Rabischong B, Botchorishvili R. Mesh-less laparoscopic treatment of apical prolapse. Facts Views Vis Obgyn. 2021 Jun;13(2):179-181. doi: 10.52054/FVVO.13.2.013. PMID 34184848